CLINICAL TRIAL: NCT03717805
Title: The Evaluation of a Preparatory Information Movie on Oocyte Aspiration: a Randomized Controlled Trial
Brief Title: The Evaluation of a Preparatory Information Movie on Oocyte Aspiration
Acronym: POAM-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: s61509
Record Dates: First submitted 2018-10-10; First posted 2018-10-24 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Infertility
Keywords: Patient-centered care; Patient information
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (1/1)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participating couples of the intervention group will receive care as usual and will watch the preparatory information movie on oocyte aspiration (POAM) 1-3 days before their oocyte aspiration. Their gynecologist or midwife will empower them to watch the movie when they call them to plan the oocyte aspiration and will send them the secured link to the movie via email.
  Interventions: Other: POAM
- Control group (No Intervention): Participating couples of the control group will receive care as usual (as will participating couples of the intervention group) and will not get access to the preparatory information movie on oocyte aspiration (POAM).

INTERVENTIONS:
Other: POAM — The new 5 minutes preparatory information movie on oocyte aspiration (POAM) details what couples can expect to happen on the day of oocyte aspiration. More specifically, it describes the patient journey detailing which procedures will happen when and how, in which room, in the presence of their partner or not, and in the presence of which healthcare professionals.
  Arms: Intervention group

SUMMARY:
The Preparatory information on Oocyte Aspiration Movie Randomized Controlled Trial (POAM-RCT) primarily aims to evaluate whether a new preparatory information on oocyte aspiration movie (POAM) decreases the anxiety of women on the day of their first oocyte aspiration for in vitro fertilisation (IVF). The control group of this RCT will receive care as usual. The intervention group will additional be given access to a preparatory information movie on oocyte aspiration 1-3 days before their oocyte aspiration via a secured link. Women's anxiety will be assessed with the 'State module of the State Trait Anxiety Inventory (STAI-state)' upon arrival at the fertility clinic on the day of the oocyte aspiration. At the same time other questionnaires will be administered. More specifically, men's anxiety and both partner's infertility specific distress will be assessed. In addition, to these secondary outcomes, clinical pregnancy with fetal heart beat and miscarriage will be followed-up 12 weeks after the oocyte aspiration. Finally, treatment delay and treatment discontinuation and long-term clinical outcomes (i.e. live birth from the first fresh embryo transfer, clinical pregnancy with fetal heart beat from the frozen embryo transfers of 1st IVF-cycle and the 12-months cumulative clinical pregnancy rates) will be followed-up twelve months after oocyte aspiration. This RCT will include 190 women (and their male partners) treated with a 1st cycle of IVF (with or without ICSI and PGD). Analysis will be according to intention to treat.

DETAILED DESCRIPTION:
Title: The evaluation of a preparatory information movie on oocyte aspiration: a Randomized Controlled Trial (POAM-RCT) Study purpose: To evaluate whether the preparatory information movie on oocyte aspiration (POAM) decreases the anxiety of ART-couples on the day of their first oocyte aspiration.

Primary outcome: The primary outcome is women's 'state anxiety', which will be assessed with the reliable 'State Trait Anxiety Inventory, state module (STAI-state)' questionnaire upon arrival at the fertility clinic on the day of the oocyte aspiration.

Secondary outcomes: Three secondary patient-reported outcomes will be assessed simultaneously with the primary outcome, upon arrival at the fertility clinic for oocyte aspiration.

First, men's state anxiety will assessed with the STAI-state questionnaire. Second and third, in both women and men, infertility-specific distress will be assessed.

The following two secondary clinical outcomes will be followed-up in all couples 12 weeks after the oocyte aspiration: clinical pregnancy with fetal heart beat and miscarriage in case of clinical pregnancy with fetal heart beat.

Other outcomes: As a follow-up the following will be extracted from the medical charts of participating couples twelve months after the oocyte aspiration: long-term clinical outcomes (i.e. live birth from the first fresh embryo transfer, clinical pregnancy with fetal heart beat from the frozen embryo transfers of 1st IVF-cycle and the 12-months cumulative clinical pregnancy rates) and long-term discontinuation parameters (i.e. censored by their medical doctor to discontinue, IVF-delay or number of untreated cycles within 12 months and IVF-discontinuation or whether or not start a 2nd IVF-cycle was started within 12 months).

Study design: Randomized controlled trial Sample size: 190 couples will be randomized to the intervention or control group Summary of eligibility criteria: Inclusion criteria: Couples treated with a 1st cycle of ART (IVF or ICSI; with or without PGD). Couples with a genetic indication for PGD can be included as they are an important patient group and are as likely as infertile patients to experience anxiety when they first come for oocyte retrieval.

Exclusion criterion: Couples going through a subsequent cycle of ART are not eligible as they are not treatment naïve, but already know, from their first cycle, what will happen on the day of oocyte aspiration.

Maximum duration of treatment of a subject: Each couple will participate from their ART-intake until the day of their first oocyte aspiration.

Couples will be asked for informed consent during their ART-intake (i.e. individual or group session with midwife; 1-3 months prior to oocyte aspiration) and will then be randomized to either the intervention group or the control group.

Participating couples of the intervention group will receive care as usual and will watch the preparatory information movie on oocyte aspiration (POAM) 1-3 days before their oocyte aspiration. Their gynecologist or midwife will empower them to watch the movie when they call them to plan the oocyte aspiration and will send them the secured link to the movie via email.

Participating couples of the control group will receive care as usual (as will participating couples of the intervention group) and will not get access to the preparatory information movie on oocyte aspiration (POAM).

When they arrive at the fertility clinic on the day of oocyte aspiration both partners of participating couples of the intervention and control group will be asked to fill out a questionnaire (5-10 minutes) before any clinical procedures are performed.

ELIGIBILITY:
Inclusion Criteria:

(i) Heterosexual woman and her partner

(ii) Dutch speaking

(iii) Treated with a 1st cycle of IVF (IVF or ICSI; with or without PGD)

Exclusion Criteria:

(i) Having already experienced an IVF-cycle in the same of another clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
Women's state anxiety | Responses on one single assessment of state-anxiety on the day of the oocyte aspiration (1-3 days after the intervention or control condition) will be compared between intervention and control group. No pre-intervention assessment, no change scores.
  Women's anxiety will be assessed with the 'State Trait Anxiety Inventory, state module (STAI-state; score 20-80, the higher the more anxious)' questionnaire (Spielberger et al, 2015; www.mingarden.com).

SECONDARY OUTCOMES:
Men's state anxiety | Responses on one single assessment of state-anxiety on the day of the oocyte aspiration (1-3 days after the intervention or control condition) will be compared between intervention and control group. No pre-intervention assessment, no change scores.
  Men's anxiety will be assessed with the 'State Trait Anxiety Inventory, state module (STAI-state; score 20-80, the higher the more anxious)' questionnaire (Spielberger et al, 2015; www.mingarden.com)
Women's infertility specific distress | Responses on one single assessment of distress on the day of the oocyte aspiration (1-3 days after the intervention or control condition) will be compared between intervention and control group. No pre-intervention assessment, no change scores.
  Women's infertility-specific distress will be assessed with the reliable 'Infertility Distress Scale (IDS; score 8-40 with the higher, the more distress)' (Pook&Krause, Fertil Steril, 2005)
Men's infertility specific stress | Responses on one single assessment of distress on the day of the oocyte aspiration (1-3 days after the intervention or control condition) will be compared between intervention and control group. No pre-intervention assessment, no change scores.
  Men's infertility-specific distress will be assessed with the reliable 'Infertility Distress Scale (IDS; score 8-40 with the higher, the more distress)' (Pook&Krause, Fertil Steril, 2005)
Clinical pregnancy with fetal heart beat | A medium duration after intervention or control condition: 12 weeks after oocyte aspiration
  A pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with a discernible heartbeat (Zegers-Hochschild et al, Hum Reprod, 2017).
Miscarriage after clinical pregnancy with fetal heart beat | A medium duration after intervention or control condition: 12 weeks after oocyte aspiration
  A miscarriage after a pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with a discernible heartbeat (Zegers-Hochschild et al, Hum Reprod, 2017).
Live birth from the first fresh embryo transfer | A long duration after intervention or control condition: One year after oocyte aspiration
  Dichotomous outcome (yes-no), which is achieved if the first fresh embryo transfer results in a live birth. More specifically, the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. Live births refer to the individual newborn; for example, a twin delivery represents two live births (Zegers-Hochschild et al, Hum Reprod, 2017).
Clinical pregnancy with fetal heart beat from the frozen embryo transfers of 1st IVF-cycle | A long duration after intervention or control condition: One year after oocyte aspiration
  Dichotomous outcome (yes-no), which is achieved if at least one clinical pregnancy with fetal heart beat is conceived after the transfer of embryos which have been frozen as a result of the first oocyte aspiration (Zegers-Hochschild et al, Hum Reprod, 2017).
12-months cumulative clinical pregnancy with fetal heart beat | A long duration after intervention or control condition: One year after oocyte aspiration
  Dichotomous outcome (yes-no), which is achieved if at least one clinical pregnancy with fetal heart beat is conceived within 12-months after oocyte aspiration
IVF-delay or number of untreated cycles within 12 months | A long duration after intervention or control condition: One year after oocyte aspiration
  The number of untreated cycles within 12 months after an unsuccessful oocyte aspiration
IVF-discontinuation | A long duration after intervention or control condition: One year after oocyte aspiration
  Dichotomous outcome (yes-no), which is achieved if a couple decides themselves (without censored by their gynaecologist) not to start a second oocyte aspiration within 12 months after their first unsuccessful oocyte aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Karen Peeraer, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- GZA Ziekenhuizen campus Sint-Augustinus, Wilrijk, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dias L, De Loecker P, Willems S, D'Hooghe TM, Vriens J, Peeraer K, Dancet EAF. A video clip detailing the patient journey on the day of oocyte retrieval in addition to the standard of care: a randomized controlled trial. Hum Reprod. 2025 Apr 1;40(4):664-674. doi: 10.1093/humrep/deaf033. PMID 40056004